CLINICAL TRIAL: NCT06085079
Title: A 24-week Two-armed Proof-of-concept Exploratory Analysis of Subcutaneous Ixekizumab Administration in Patients With Recalcitrant Non-infectious Intermediate, Posterior, Panuveitis, or Chronic Steroid-dependent Anterior Uveitis.
Brief Title: Ixekizumab for the Management of Refractory Non-Infectious Uveitis: A Proof-of-Concept Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts Eye Research and Surgery Institution (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IXE-1001
Record Dates: First submitted 2023-04-03; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate; Panuveitis
MeSH Terms: conditions — Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate; Panuveitis

STUDY DESIGN:
Intervention Model Description: Arm 1: Subjects will self-administer subcutaneous injection of ixekizumab during the baseline week (Week 0) using a loading dose of 160 mg of subcutaneous ixekizumab (Taltz), followed by 80 mg of subcutaneous ixekizumab Q2 weeks for 24-weeks.
  Arm 2: Subjects will self-administer subcutaneous injection of ixekizumab during the baseline week (Week 0) using a loading dose of 160 mg of subcutaneous ixekizumab (Taltz), followed by 80 mg of subcutaneous ixekizumab Q4 weeks for 24-weeks.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2-week dosing (Experimental): Subjects will self-administer subcutaneous injection of ixekizumab during the baseline week (Week 0) using a loading dose of 160 mg of subcutaneous ixekizumab (Taltz), followed by 80 mg of subcutaneous ixekizumab Q2 weeks for 24-weeks.
  Interventions: Drug: Ixekizumab Prefilled Syringe
- 4-week dosing (Experimental): Subjects will self-administer subcutaneous injection of ixekizumab during the baseline week (Week 0) using a loading dose of 160 mg of subcutaneous ixekizumab (Taltz), followed by 80 mg of subcutaneous ixekizumab Q4 weeks for 24-weeks.
  Interventions: Drug: Ixekizumab Prefilled Syringe

INTERVENTIONS:
Drug: Ixekizumab Prefilled Syringe — Ixekizumab is a humanized IgG4 monoclonal antibody that binds with high affinity and specificity to IL-17A. This medication is currently approved for the treatment of plaque Ps, ankylosing spondylitis, and psoriatic arthritis.

SUMMARY:
The objective of this study is to explore the efficacy of ixekizumab in treating patients with a diagnosis of non-infectious intermediate, posterior, panuveitis, or chronic steroid-dependent anterior uveitis who had failed treatment with a classic synthetic DMARD including methotrexate, mycophenolate, cyclosporin, azathioprine, cyclophosphamide and/or at least one anti-TNF agent including adalimumab, infliximab, etanercept, golimumab or certolizumab.

DETAILED DESCRIPTION:
This is a 24-week open label analysis of subcutaneous ixekizumab (taltz) in patients with non-infectious intermediate, posterior, panuveitis, and chronic steroid-dependent anterior uveitis. The study visits are held at Massachusetts Eye Research and Surgery Institution (MERSI) in Waltham, Massachusetts. The study is aiming to enroll 20 subjects. This is a two-armed study in which Group A receives ixekizumab every 2 weeks and Group B receives ixekizumab every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Diagnosis of non-infectious intermediate, posterior, panuveitis, or chronic steroid dependent anterior uveitis
3. Failure of at least one classic synthetic DMARD including Methotrexate, Mycophenolate, Cyclosporin, Azathioprine, Cyclophosphamide, and/or at least one anti-TNF agent including Adalimumab, Infliximab, Etanercept, Golimumab or Certolizumab
4. Active disease at screening visit
5. At least 1 of the following parameters in at least one eye:

   * active inflammatory chorioretinal and/or inflammatory retinal vascular lesions
   * ≥ 1+ vitreous haze (Nussenblatt criteria)
   * ≥ 2+ anterior chamber cells (National Eye Institute/Standardization of Uveitis Nomenclature criteria)
   * Cystoid macular edema, seen on optical coherence tomography and/or fluorescein angiography
   * FA leakage pattern deemed by investigators to be suggestive of active intermediate, posterior, and panuveitis, including optic disc, retinal vascular, and macular leakages
   * Active snowbanking

Exclusion Criteria:

* The presence of only acute anterior uveitis.
* Serpiginous choroidopathy
* Subject with prior inadequate response to high-dose oral corticosteroids (> 60 mg of prednisone)
* Subject with confirmed or suspected infectious uveitis
* Patients with intraocular pressure of ≥ 25 mmHg or evidence of optic nerve injury
* Corneal or lens opacity that precludes adequate ophthalmic evaluation.
* Patients likely to undergo cataract surgery during the duration of the trial.
* Patients with Best Corrected Visual Acuity (BCVA) less than 20 letters (Early Treatment Diabetic Retinopathy Study)
* Dose of concomitant immunosuppressive therapy at the baseline visit:

  * Methotrexate (MTX) ˃ 25 mg per week
  * Cyclosporine ˃ 4 mg/kg per day
  * Mycophenolate mofetil ˃ 3 grams per day or an equivalent drug to mycophenolate mofetil (e.g. mycophenolic acid) at an equivalent dose approved by the medical monitor.
  * Azathioprine ˃ 175 mg per day
  * Tacrolimus (oral formulation) > 8 mg per day
* If entering the study on 1 concomitant immunosuppressive therapy, dose has been increased within the last 28 days prior to Baseline visit.
* Subject has received Retisert® (implant) within 3 years prior to the Baseline visit or that has had complications related to the device. Subject has had Retisert® (implant) removed within 90 days prior to the Baseline visit or has had complications related to the removal of the device
* Subject has received intraocular or periocular corticosteroids within 30 days prior to Baseline visit
* Subject with proliferative or severe non-proliferative diabetic retinopathy or clinically significant macular edema due to diabetic retinopathy
* Subject with neovascular/wet age-related macular degeneration
* Subject with abnormality of vitreo-retinal interface (i.e., vitreomacular traction, epiretinal membranes, etc.) with the potential for macular structural damage independent of the inflammatory process, deemed macular pathology is deemed by a retinal specialist to be a potential cofounder of patient's visual acuity reduction
* Subject with severe vitreous haze that precludes visualization of the fundus at the baseline visit
* Subject has received Ozurdex® (dexamethasone implant) within 6 months prior to the baseline visit
* Subject has received intravitreal anti-VEGF therapy within 45 days of the Baseline visit for Lucentis® (ranibizumab) or Avastin® (bevacizumab) or within 60 days of the Baseline visit for anti-VEGF Trap (aflibercept)
* Subject has received intravitreal methotrexate within 90 days prior to the Baseline visit
* Subject on systemic carbonic anhydrase inhibitor within 1 week prior to Screening visit
* Subject with macular edema as the only sign of uveitis
* Subject with a history of scleritis
* Subject with intolerance to high-dose oral corticosteroids (equivalent of oral prednisone 1 mg/kg/day or 60 to 80 mg/day)
* Subject on cyclophosphamide within 30 days prior to the Baseline visit
* Participation in other investigational drug or device clinical trials within 30 days prior to Day 0 or planning to participate in other investigational drug or device clinical trials within 180 days following 48 weeks after day 0. This includes both ocular and non-ocular clinical trials
* Major surgery within 8 weeks prior to screening or planned major surgery within 6 months following randomization
* Treatment with intravenous gamma globulin or plasmapheresis during the course of the trial
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline
* History of severe allergic or anaphylactic reactions to human, humanized monoclonal antibodies
* Prior history of Crohn's Colitis or Ulcerative Colitis
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, liver disease or peptic ulcer disease)
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds)
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Active tuberculosis (TB) requiring treatment within the previous 3 years. Patients should be screened for latent TB and, if positive, treated following local practice guidelines prior to initiating trial. Patients treated for tuberculosis with no recurrence in 3 years are permitted
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of active malignant disease, malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured)
* Pregnant women or breast-feeding mothers
* Patients with reproductive potential not willing to use an effective method of contraception
* History of alcohol, drug, or chemical abuse within 1 year prior to screening.
* Serum creatinine > 1.6 mg/dL (141 μmol/L) in female patients and > 1.9 mg/dL (168 μmol/L) in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN)
* Total Bilirubin > 1.5 ULN
* Platelet count < 100 x 109/L (100,000/mm3)
* Hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L)
* White Blood Cells < 3.0 x 109/L (3000/mm3)
* Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3)
* Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
* Positive Hepatitis BsAg, or Hepatitis C antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Assessed around week 10
  The four components of the composite endpoint will each be graded dichotomously (i.e., yes, or no for success), and include visual acuity, control of inflammation, tapering of medication therapy, and reduction of cystoid macular edema. Clinical response will be defined by improvement in at least one parameter with worsening in none, and well controlled intraocular inflammation.

SECONDARY OUTCOMES:
Intraocular pressure | This will be measured and assessed throughout the entire 24-week study period up until the patient's final visit.
  Intraocular pressure is a number between 0 and 100 mmHg, with most values ranging from 5-30 and normal of 10-21.
Subjective Visual Benefit | This will be measured and assessed throughout the entire 24-week study period up until the patient's final visit.
  The National Eye Institute Visual Functioning Questionnaire - 25 (VFQ-25) will measure the patient's assessment of his or her vision and problems and how these problems impact their quality of life. Responses are quantified numerically for each section. These responses have specific ranges: 1 to 6 for "General Health and Vision" (section 1, with lower number response signifying better health outcomes); 1 to 6 for "Difficulties with Activities" (section 2, with lower number response signifying less difficulty with activities); 1-5 for "Responses to Vision Problems" (section 3, with lower number response signifying more negative responses to vision problems).
Adverse Event frequency | This will be monitored and assessed throughout the entirety of the 24-week study period and through 30 days following the last administration of study treatment.
  The following safety endpoints will be measured: allergic reactions, hypersensitivity, malignancies, infections (upper respiratory tract, urinary tract, sinusitis, tonsillitis, bronchitis, cystitis), serious infections, candidiasis, MACE, Crohn's disease, ulcerative colitis, injection site reactions (mild, moderate, severe), diarrhea, depression, muscle spasm, hypertension, osteoarthritis, psoriatic arthritis, fatigue, headache, back pain, LFT elevation, lipid elevation, cerebro-cardiovascular events, depression/suicide, death. The development or worsening of any medical problems will be documented through adverse event monitoring at each study visit. The frequency of each adverse event across all subjects will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: C. Stephen Foster, MD, FACS, FACR, Principal Investigator — Founder of research site
Locations (1):
- Massachusetts Eye Research and Surgery Institution, Waltham, Massachusetts, United States